CLINICAL TRIAL: NCT01110018
Title: A Single-centre, Open-label, Sequential, Cross-over Study to Examine the Safety, Tolerability and Pharmacokinetics of 3 Ascending Single Intravenous Doses, a Single 1000μg Oral Dose and a Single 1000μg Inhaled Dose of GSK573719 in Healthy Male Volunteers.
Brief Title: GSK573719 IV Enabling Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112008
Record Dates: First submitted 2010-04-15; First posted 2010-04-23 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Tolerability; COPD; Safety; Muscarinic receptor (mAChR) antagonist; GSK573719; Healthy subjects; Pharmacokinetics; IV study
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — GSK573719; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Period 1 (Active Comparator): 20μg intravenous infusion administered over 30 minutes
  Interventions: Drug: GSK573719 (SOLUTION)
- Period 2 (Active Comparator): 1000μg Oral dose
  Interventions: Drug: GSK573719 (SOLUTION)
- Period 3 (Active Comparator): 50μg Intravenous infusion administered over 30 minutes
  Interventions: Drug: GSK573719 (SOLUTION)
- Period 4 (Active Comparator): 1000μg Inhaled dose
  Interventions: Drug: GSK573719 (INHALATION POWDER)
- Period 5 (Active Comparator): 100μg Intravenous infusion administered over 30 minutes
  Interventions: Drug: GSK573719 (SOLUTION)

INTERVENTIONS:
Drug: GSK573719 (SOLUTION) — 20μg /mL solution for IV and Oral dosing
  Arms: Period 1; Period 2; Period 3; Period 5
Drug: GSK573719 (INHALATION POWDER) — 500μg inhalation powder delivered via Novel Dry Powder Inhaler. GSK573719 1000μg per dose (2x 500μg strips in device).
  Arms: Period 4

SUMMARY:
A single-centre, open-label, sequential, cross-over study to examine the safety, tolerability and pharmacokinetics of 3 ascending single intravenous doses, a single 1000μg oral dose and a single 1000μg inhaled dose of GSK573719 in healthy male volunteers.

DETAILED DESCRIPTION:
GSK573719 is a high-affinity, specific, reversible muscarinic receptor (mAChR) antagonist which is being developed for the treatment of Chronic Obstructive Pulmonary Disease (COPD). The long duration of action of GSK573719, when administered via inhalation to humans, supports the potential for use as a long acting bronchodilator for COPD.

This will be an open-label, single dose, dose-ascending study in healthy male subjects to establish well tolerated intravenous (IV) dose of GSK573719 to be administered in a subsequent definitive human radiolabel metabolic study. The pharmacokinetics and the bioavailability of a single oral and a single inhaled dose of GSK573719 will also be evaluated.

Blood and urine samples for pharmacokinetic analysis will be taken at regular intervals up to 48 hours after dosing. Safety will be assessed by measurement of heart rate, blood pressure, ECG, lead II monitoring and twenty four hour Holter monitoring, safety laboratory data and review of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until follow up.
* Body Mass Index within the range 18-30 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Average QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.
* Non-smokers (never smoked or not smoking for >6 months with <10 pack years history (Pack Years = (cigarettes per day smoked/20) x number of years smoked)

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-04-28 (Actual); Primary Completion 2010-06-09 (Actual); Study Completion 2010-06-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of GSK573719 | Study duration (5 weeks)

SECONDARY OUTCOMES:
IV dose plasma PK parameters: AUC(0-∞) (if calculable), AUC(0-t), and Cmax, tlast, CL, Vss, MRT, λz and t½ | Pre-dose to 24h post-dose (48h post-dose in IV dose 3)
Oral and Inhaled dose plasma PK parameters: AUC(0-∞) (if calculable), AUC(0-t) and Cmax, tmax, tlast, F, λz and t½, if calculable. | Pre-dose to 24h post-dose
Urine PK parameters for all routes of administration: CLr, t½, Ae(0-2), Ae(0-4) , Ae(0-8) , Ae(0-12) , Ae(0-24) , Ae(0-36), Ae(0-48), fe, F , AUER(0-18), AUER(0-36) if available, AUER(0-∞). | 0-48h post-dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 112008 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112008?search=study&study_ids=112008#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 112008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register